CLINICAL TRIAL: NCT05374850
Title: Impact of Cervical Sagittal Parameters on Interlaminar Epidural Steroid Injection Treatment Outcomes in Patients With Cervical Disc Herniation
Brief Title: Impact of Cervical Parameters to Interlaminar Epidural Steroid Injection Treatment Outcomes in Patients With Cervical Disc Herniation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 07.01.2022.82
Record Dates: First submitted 2022-04-20; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Cervical Disc Herniation
Keywords: cervical sagittal parameters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cervical Interlaminar Epidural Steroid Injection — This intervention is applied mostly for cervical disc herniation.The intervention was carried out under sterile conditions with the C-arm fluoroscopy guidance. It is performed via spinal needle and the needle is inserted into the epidural space, then combined local anesthetics and glucocorticoids is delivered to the epidural space.

SUMMARY:
This study is aim to disclose the effect of cervical parameters, whether they change the outcomes of epidural steroid injection treatment in patients with cervical disc herniation. The patients who had cervical disc herniation and had been performed interlaminar epidural steroid injection were included. We hypothesized that participants with abnormal cervical spine alignment parameters were less likely to benefit from treatment.

DETAILED DESCRIPTION:
The objective of this study is to reveal the impact of cervical sagittal parameters on interlaminar epidural steroid injections in patients with cervical disc herniation. Patients who have suffered from cervical radicular pain for at least 3 months and been diagnosed with cervical radiculopathy in our pain clinic in the subsequent stage, with a clinical and physical examination, as well as radiologic assessments, were included in the study. Other inclusion criteria were intractable pain over the neck despite conservative treatment and being between the ages of 18 and 65. Patients with a history of epidural steroid injections carried out in the previous 3 months, patients with a history of cervical spine surgery, patients with systemic and/or local infections, malignancy, bleeding diathesis, acute fracture, known allergy to contrast material and/or local anesthetic substances, known history of any psychiatric disorder, and patients with a history of pregnancy were excluded from the study. Verbal and written informed consent was obtained from all patients participating in the study.

In addition to the recording of the demographic data of the patients participating in this study (age, sex, duration of symptoms, etc.), their sagittal parameters angles (C2-C7 cervical lordosis, C2-C7 sagittal vertical axis, C7 slope and spino-cranial angle) and the numeric rating scale (NRS) was employed before the procedure and in the 1st hour, 3rd week, and 3rd month after the procedure. Short Form-12 Health Survey (SF-12) was employed before the procedure and in the 3rd week and 3rd month after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suffered from neck pain for at least 3 months and been diagnosed with cervical radiculopathy
* Intractable pain despite conservative treatment and being between the ages of 18 and 65
* Patients who will be performing with an interlaminar epidural steroid injection(ILESI)

Exclusion Criteria:

* Patients with a history of ILESI carried out in the previous 3 months,
* Patients with a history of cervical surgery,
* Patients with systemic and/or local infections,
* Malignancy,
* Bleeding diathesis,
* Acute fracture,
* Known allergy to contrast material and/or local anesthetic substances,
* Known history of any psychiatric disorder
* Patients with a history of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ,between the ages of 18 and 65, who diagnosed with cervical radiculopathy due to disc herniation in our pain clinic and who are resistant to conservative treatment, so the patients to be treated with ILESI procedure.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Change of pain severity from baseline to each checkpoints from pre-interventional time to post-interventional 1st hour, 3rd week and 3rd month
  A numeric (or numerical) scale, also known as a Numerical Rating Scale (NRS), is basically any scale that renders a quantitative symbolization of an attribute. This type of scale is used by presenting the respondent with an ordered set from which to choose, for example, 1 to 10, coupled with anchors. These anchors can be put at the endpoints or at each point on the scale.

SECONDARY OUTCOMES:
Short-form 12(SF-12) | Change of life quality from baseline to each checkpoints from pre-interventional time to post-interventional 3rd week and 3rd month
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
The Neck Disability Index (NDI) | Change of functionality from baseline to each checkpoints from baseline to each checkpoints from pre-interventional time to post-interventional 3rd week and 3rd month
  Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.

CONTACTS AND LOCATIONS:
Overall Officials: SAVAS SENCAN, Principal Investigator — Marmara University Pendik Training and Research Hospital
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mesregah MK, Feng W, Huang WH, Chen WC, Yoshida B, Mecum A, Mandalia K, Van Halm-Lutterodt N. Clinical Effectiveness of Interlaminar Epidural Injections of Local Anesthetic with or without Steroids for Managing Chronic Neck Pain: A Systematic Review and Meta-Analysis. Pain Physician. 2020 Jul;23(4):335-348. PMID 32709169
- [Background] Manchikanti L, Knezevic NN, Navani A, Christo PJ, Limerick G, Calodney AK, Grider J, Harned ME, Cintron L, Gharibo CG, Shah S, Nampiaparampil DE, Candido KD, Soin A, Kaye AD, Kosanovic R, Magee TR, Beall DP, Atluri S, Gupta M, Helm Ii S, Wargo BW, Diwan S, Aydin SM, Boswell MV, Haney BW, Albers SL, Latchaw R, Abd-Elsayed A, Conn A, Hansen H, Simopoulos TT, Swicegood JR, Bryce DA, Singh V, Abdi S, Bakshi S, Buenaventura RM, Cabaret JA, Jameson J, Jha S, Kaye AM, Pasupuleti R, Rajput K, Sanapati MR, Sehgal N, Trescot AM, Racz GB, Gupta S, Sharma ML, Grami V, Parr AT, Knezevic E, Datta S, Patel KG, Tracy DH, Cordner HJ, Snook LT, Benyamin RM, Hirsch JA. Epidural Interventions in the Management of Chronic Spinal Pain: American Society of Interventional Pain Physicians (ASIPP) Comprehensive Evidence-Based Guidelines. Pain Physician. 2021 Jan;24(S1):S27-S208. PMID 33492918
- [Background] Azimi P, Yazdanian T, Benzel EC, Hai Y, Montazeri A. Sagittal balance of the cervical spine: a systematic review and meta-analysis. Eur Spine J. 2021 Jun;30(6):1411-1439. doi: 10.1007/s00586-021-06825-0. Epub 2021 Mar 27. PMID 33772659
- [Background] Iyer S, Nemani VM, Nguyen J, Elysee J, Burapachaisri A, Ames CP, Kim HJ. Impact of Cervical Sagittal Alignment Parameters on Neck Disability. Spine (Phila Pa 1976). 2016 Mar;41(5):371-7. doi: 10.1097/BRS.0000000000001221. PMID 26571157
- [Background] Nicholson KJ, Millhouse PW, Pflug E, Woods B, Schroeder GD, Anderson DG, Hilibrand AS, Kepler CK, Kurd MF, Rihn JA, Vaccaro A, Radcliff KE. Cervical Sagittal Range of Motion as a Predictor of Symptom Severity in Cervical Spondylotic Myelopathy. Spine (Phila Pa 1976). 2018 Jul 1;43(13):883-889. doi: 10.1097/BRS.0000000000002478. PMID 29095412